CLINICAL TRIAL: NCT06684314
Title: PROphylactic Efanesoctocog Alfa Therapy Evaluated for Critical Joint Health in Hemophilia A Treatment: The PROTECT-ALT Study
Brief Title: A Study to Evaluate Impact of Efanesoctocog Alfa on Long-term Joint Health in Participants With Hemophilia A in Taiwan
Acronym: PROTECT-ALT
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18067; U1111-1308-9835 (Registry Identifier: WHO ICTRP)
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Hemophilia A
Keywords: Classic Hemophilia; Factor VIII Deficiency; Haemophilia; Hemophilia; Hemarthrosis; Blood Coagulation Disorders, Inherited; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn
MeSH Terms: conditions — Hemophilia A; Hemarthrosis; Blood Coagulation Disorders, Inherited; Hematologic Diseases; Coagulation Protein Disorders; Hemorrhagic Disorders; Genetic Diseases, Inborn | interventions — BIVV001

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Efanesoctocog alfa: Participants observed receiving treatment with efanesoctocog alfa for hemophilia A
  Interventions: Drug: Efanesoctocog alfa

INTERVENTIONS:
Drug: Efanesoctocog alfa — This study will not administer any treatment, only observe the treatment as prescribed in real-world clinical practices.
  Other Names: ALTUVIIIO; BIVV001

SUMMARY:
This is a national, multicenter, retrospective/prospective, observational study in Taiwan designed to assess effectiveness, safety, and usage of efanesoctocog alfa prophylaxis treatment in hemophilia A participants. The data related to efanesoctocog alfa effectiveness, safety and usage will be recorded prospectively during routine visits for up to 5 years following enrollment initiation and the retrospective data will be collected at least 12 months and up to 24 months prior to efanesoctocog alfa initiation. Joint imaging data will be collected in centers performing Joint U/S and/or MRI (≥6 years old). At least 12 months of retrospective data will also be collected from medical records, as available. Prospectively collected data will be recorded at routine clinical visits during a five-year follow-up period. The end of study is defined as the last participant's last visit. No intervention will be administered, and no study related visits are required.

ELIGIBILITY:
Inclusion Criteria:

* Participants with all ages and diagnosis of moderate-severe hemophilia A without current and/or at least three years of un-detectable inhibitor (<0.6 BU)
* Participants with moderate to severe hemophilia A as defined by FVIII level ≤ 5%
* Participants starting efanesoctocog alfa prophylaxis treatment as per standard of care no more than three months prior to the enrollment date
* Participants aged 6 years and older are able to undergo MRI examinations (sedation given, if necessary, and per investigator discretion)
* Participants are able to undergo joint examinations
* Physician's decision to treat the participant with efanesoctocog alfa is made prior to and independently of participation in the study
* Signed and dated informed consent provided by the participant, or by the participant's legally acceptable representative for participants under the legal age before any study-related activities are undertaken. Assent should be obtained for pediatric participants according to local regulations

Exclusion Criteria:

* Participants with coagulation disorders other than hemophilia A
* Participants diagnosed with other known bleeding disorder
* Participants currently receive factor therapy and have signs of decreased response to FVIII therapy
* Participants with a baseline Radiological Pettersson score (PS) of greater than 6 for each individual ankle
* Enrollment in another concurrent clinical interventional study, or intake of an Investigational Medicinal Product within 3 months prior to inclusion in this study
* Pregnant female participants

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants from medical centers in Taiwan will be enrolled in the study after the introduction of efanesoctocog alfa for the treatment of hemophilia A. Eligible participants will include all ages, sexes and moderate to severe hemophilia A severities under efanesoctocog alfa prophylaxis treatment and able to undergo joint and/or MRI examinations during routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2031-08-28 (Estimated); Study Completion 2031-08-28 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in total scores of the Hemophilia Joint Health Score (HJHS) for all joints | At 1, 2, 3, 4 and 5 years
  The HJHS summarizes joint health by providing a clinical score in the domain of body structure and function (i.e., impairment), of the joints most commonly affected by bleeding in hemophilia: (left ankle, right ankle, left elbow, right elbow, left knee, right knee). The HJHS consists of assessments of swelling, duration of swelling, muscle atrophy, crepitus on motion, flexion loss, extension loss, joint pain and strength for elbows, knees and ankles and a global gait score. A higher score indicates worse joint health.
Change from baseline in annualized joint bleeding rate (AjBR) for treated and untreated bleeds | At 1, 2, 3, 4 and 5 years
  The AjBR is defined as the number of joint bleeding episodes occurring during the treatment period divided by the duration of the treatment period in days multiplied by 365.25. All types of joint bleeding episodes (spontaneous, traumatic, and type unknown) will be included in determining the annualized number.
Number of target joint development, resolution and/or recurrence | At 1, 2 ,3, 4 and 5 years

SECONDARY OUTCOMES:
Annualized bleeding rate (ABR) by type and location for treated and all (treated and untreated) bleeds | At 1, 2, 3, 4 and 5 years
ABR for all bleeding episodes, including untreated bleeding episodes | At 1, 2, 3, 4 and 5 years
Percentage of participants with zero joint bleeds | At 1, 2, 3, 4 and 5 years
Percentage of bleeding episodes treated with a single injection of efanesoctocog alfa | At 1, 2, 3, 4 and 5 years
Number of injections and doses of efanesoctocog alfa to treat a bleeding episode | At 1, 2, 3, 4 and 5 years
Annualized factor consumption per participant (IU/kg) assessed by prescription during the follow-up period | At 1, 2, 3, 4 and 5 years
Annualized injection frequency per participant (assessed by prescription) during the followup period | At 1, 2, 3, 4 and 5 years
Treatment adherence (%) as judged by the physician during the follow-up period | At 1, 2, 3, 4 and 5 years
Occurrence of a change in treatment regimen at baseline and follow-up | 5 years
Change from baseline in Hemophilia Early Arthropathy Detection with Ultrasound (HEAD-US) total/domain scores in all joints | Every 6 months for 5 years
Change from baseline in joint status on functional HJHS | At 1, 2, 3, 4 and 5 years
Number and percentage of joints with no prior joint damage at baseline, without joint damage on joint ultrasound | At 5 years
Changes from baseline in HEAD-US synovitis domain | Every 6 months for 5 years
Change from baseline in MRI score | At 1, 2, 3, 4 and 5 years
Number and percentage of participants without joint damage on MRI | At 1, 2, 3, 4 and 5 years
Number and percentage of joints with no prior joint damage at baseline, without joint damage on MRI | At 1, 2, 3, 4 and 5 years
Hemostatic response/physician reported during peri-operative period for surgery (major, minor) with efanesoctocog alfa | 5 years
Number of injections and dose per injection required to maintain hemostasis during perioperative period for surgery (major, minor) | 5 years
Total efanesoctocog alfa consumption (IU) during perioperative period for surgery (major, minor) | 5 years
Number and type of blood component transfusions used during perioperative period for surgery | 5 years
Estimated blood loss (mL) during perioperative period for major surgery | 5 years
Number of transfusions required for surgery (intraoperative and post-operative period) | 5 years
Duration of hospitalization (major, minor) | 5 years
Occurrence of adverse events (AEs), serious adverse events (SAEs) and adverse events of special interest (AESI) | 5 years
Development of inhibitors (neutralizing antibodies directed against factor FVIII as determined via the Nijmegen modified Bethesda assay) | 5 years
Change from baseline in HAL (haemophilia activities list) for adult participants only | At 1, 2, 3, 4 and 5 years
  HAL contains 42 items across 7 domains: lying down/ sitting/ kneeling/ standing, functions of the legs, functions of the arms, use of transportation, self-care, household tasks and leisure activities and sports. Items are scored on a 6-point Likert scale ('impossible', 'always', 'usually', 'sometimes', 'almost never', 'never'), with a 'not applicable' option for some items. A summary score as well as component scores (upper extremity, basic lower extremity and complex lower extremity) can be calculated. The scores are converted to a normalized score from 0 to 100, where higher scores represent a better functional status.
Change from baseline in PROMIS pain intensity 3a questionnaire for adult participants only | At 1, 2, 3, 4 and 5 years
  The PROMIS Pain Intensity instrument assesses how much a person hurts. The Pain Intensity short forms are universal rather than disease specific. The 1a and the first two items within the PROMIS Scale- Pain Intensity 3a short form assesses pain intensity over the past seven days. The version 2.0 of Pain Intensity 3a instruments are available for adults (ages 18+), and the version v1.0 of Pediatric Pain Intensity 1a self-report (ages 8-17) will be used for this study.
Change from baseline in PROBE full questionnaire for adult participants only | At 1, 2, 3, 4 and 5 years
  The PROBE questionnaire assesses participant reported outcomes in people with hemophilia and people without a bleeding disorder. The PROBE questionnaire is comprised of four major sections, including demographic data, general health problems, hemophilia-related health problems and health-related quality of life. It combines generic and disease-specific outcomes in 29 questions.
Change from baseline in Ped-HAL (haemophilia activities list) for adolescent participants only (≥ 12 to <18 years) | At 1, 2, 3, 4 and 5 years
  PedHAL contains 53 items across 7 domains: sitting/ kneeling/ standing, functions of the legs, functions of the arms, use of transportation, self-care, household tasks and leisure activities and sports. It consists of a participant version (8-18 years) and parent version (4-17 years). Items are scored on a 6-point Likert scale ('impossible', 'always', 'usually', 'sometimes', 'almost never', 'never'), with a 'not applicable (N/A)' scoring option for all items. A summary score as well as domain scores can be calculated. The scores are converted to a normalized score from 0 to 100, where higher scores represent a better functional status.
Change from baseline in PROMIS pain intensity 1a questionnaire for adolescent participants only (≥ 12 to <18 years) | At 1, 2, 3, 4 and 5 years
  The PROMIS Pain Intensity instrument assesses how much a person hurts. The Pain Intensity short forms are universal rather than disease specific. The 1a and the first two items within the PROMIS Scale- Pain Intensity 3a short form assesses pain intensity over the past seven days. The version 2.0 of Pain Intensity 3a instruments are available for adults (ages 18+), and the version v1.0 of Pediatric Pain Intensity 1a self-report (ages 8-17) will be used for this study.
Change from baseline in PROBE full questionnaire for adolescent participants only (≥ 12 to <18 years) | At 1, 2, 3, 4 and 5 years
  The PROBE questionnaire assesses participant reported outcomes in people with hemophilia and people without a bleeding disorder. The PROBE questionnaire is comprised of four major sections, including demographic data, general health problems, hemophilia-related health problems and health-related quality of life. It combines generic and disease-specific outcomes in 29 questions.
Change from baseline in Ped-HAL (pediatric haemophilia activities list) for pediatric participants only (12 years and younger) | At 1, 2, 3, 4 and 5 years
  PedHAL contains 53 items across 7 domains: sitting/ kneeling/ standing, functions of the legs, functions of the arms, use of transportation, self-care, household tasks and leisure activities and sports. It consists of a participant version (8-18 years) and parent version (4-17 years). Items are scored on a 6-point Likert scale ('impossible', 'always', 'usually', 'sometimes', 'almost never', 'never'), with a 'not applicable (N/A)' scoring option for all items. A summary score as well as domain scores can be calculated. The scores are converted to a normalized score from 0 to 100, where higher scores represent a better functional status.
Number of hospitalizations excluding surgery and admission/discharge diagnoses | Change from baseline at 1, 2, 3, 4 and 5 years
Number of hospitalization days | Change from baseline at 1, 2, 3, 4 and 5 years
Number of intensive care unit (ICU) stays | Change from baseline at 1, 2, 3, 4 and 5 years
Number of emergency room visits | Change from baseline at 1, 2, 3, 4 and 5 years
Number of outpatient visits | Change from baseline at 1, 2, 3, 4 and 5 years

CONTACTS AND LOCATIONS:
Locations (10):
- Taiwan (10):
  - Investigational Site Number : 1580008, Changhua
  - Investigational Site Number : 1580009, Kaohsiung City
  - Investigational Site Number : 1580010, Kaohsiung City
  - Investigational Site Number : 1580005, Taichung
  - Investigational Site Number : 1580006, Taichung
  - Investigational Site Number : 1580007, Taichung
  - Investigational Site Number : 1580001, Taipei
  - Investigational Site Number : 1580003, Taipei
  - Investigational Site Number : 1580002, Taipei
  - Investigational Site Number : 1580004, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org